CLINICAL TRIAL: NCT06131268
Title: The Role of Negr1 In Modulating Neuroplasticity in Major Depression (RONIN)
Acronym: RONIN
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RONIN
Record Dates: First submitted 2023-04-13; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-08

CONDITIONS: Major Depressive Disorder; Bipolar Affective Disorder, Currently Depressed, Moderate
Keywords: major depressive disorder; NEGR1 protein; antidepressants; venlafaxina; NEGR1 mRna; brain connectivity
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Lymphoma, Follicular | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with Major Depression (Group 1) (Experimental): They will be evaluated at baseline (T0) and at 4 weeks from the setting of drug treatment with venlafaxine (T1)
  Interventions: Drug: Venlafaxine
- Bipolar disorder patients (Group 2) (No Intervention): Venlafaxine will not be administered. They will be valuated both at T0 and after 4 weeks (T1).
- Healthy controls (Group 3) (No Intervention): Venlafaxine will not be administered. They will be evaluated only at baseline (T0).

INTERVENTIONS:
Drug: Venlafaxine — we will recruit a cohort of 10 MDD patients currently receiving evidence-based treatments for depression (including treatment with an antidepressant drug such as SSRIs/SNRIs) who will be switched to the antidepressant venlafaxine and followed along for 4 weeks (Group 1). The switch from the ongoing treatment to venlafaxine will must be required by therapeutical needs (null or partial response and/or poor tolerability or compliance to ongoing therapy) according to the indications of the principle clinical guidelines for the treatment of MDD and it is independent of the decision of including the patient in the study.
  Arms: Patients with Major Depression (Group 1)

SUMMARY:
Patients belonging to Group 1 (Major Depression) and 2 (Bipolar Disorder) will be tested with psychometric and functional scales at baseline (T0) and after 4 weeks of pharmacological therapy (T1), to evaluate clinical and functional response to treatment. MDD patients will be screened for the lifetime and recent occurrence of clinically meaningful suicidal ideation and behavior prior to recruitment (-T1). Moreover, in the MDD group, the emergence of clinically meaningful suicidal ideation and behavior will be evaluated at the baseline (T0) and after 4 weeks (T1) by means of the C-SSRS, accordingly to the routine clinical practice. Furtherly, to accomplish the pursues of this research, the two groups will undergo neuroimaging evaluation and a blood collection at the two timepoints for measuring the expression of ncRNA before and after treatment. Meanwhile, a lumbar puncture (LP) for CSF collection will be carried out at the baseline, measuring central levels of Negr-1 and other biomarkers of neurotropism potentially related to the aforementioned role of Negr1 in MDD. Group 3 will be comprehensive of 10 subjects without current or previous diagnosis of psychiatric disorders (healthy controls), who will be evaluated at baseline with psychometric and functional scales, neuroimaging and blood samples collection for ncRNA. Data obtained by the multimodal assessment of HCs at the baseline will be employed as normalization features in the statistical analysis of patients' data.

DETAILED DESCRIPTION:
In this clinical trial, the investigators will recruit a cohort consisting of 10 patients with MDD who will be evaluated at baseline (T0) and at 4 weeks from the setting of drug treatment with venlafaxine (T1). The sample consists of patients already being treated with antidepressant drugs (e.g., drugs SSRI/SNRIs) for whom it was necessary to switch to venlafaxine therapy medication due to poor/no response or poor tolerability to current therapy according to the indications of the major clinical guidelines for the treatment of MDD and completely independently of study participation.

To distinguish clinical variations related to the clinical course of depression, the investigators will also recruit a cohort of 10 patients with bipolar disorder, suffering from a current depressive episode (Group 2) and who will be assessed both at T0 and after 4 weeks (T1). To identify markers blood and neuroimaging markers of MDD, will be recruited 10 healthy controls without current psychiatric history (Group 3), who will be evaluated only at baseline (T0). After signing informed consent and recruitment, demographic data (age, sex, level of education, etc.) and clinical data (past and current diagnoses, comorbidities, habits smoking, past therapy, age at onset, etc.) were collected from patients and healthy controls, as possible variables confounders to the clinical course of MDD. Patients with MDD and bipolar disorder will be tested with psychometric and functional scales (BPRS, MADRS, HDRS, GAF) at baseline (T0) and after 4 weeks of therapy (T1), to assess the change in clinical picture.

The presence or occurrence of suicidal ideation or behavior in patients with MDD will be assessed by clinical interview and administration of the C-SSRS at baseline (T0) and after 4 weeks of therapy (T1). (In addition, the three groups at baseline will perform structural and functional brain MRI associated with EEG and the collection of two peripheral venous blood samples. All assessments will be repeated at T1 (at 4 weeks) for Groups 1 and 2 of MDD and DB patients. More over, at baseline, patients in Group 1 and 2 will undergo spinal tap (PL), with collection of a sample of fluid cerebrospinal fluid, for measurement of central levels of Negr-1 and other biomarkers of neurotropism potentially involved in Negr1 activity in MDD. In the cerebrospinal fluid and peripheral blood biological samples, obtained from the three groups of subjects, the levels of gene expression (mRNA) and protein levels of Negr-1 and other biomarkers involved in the modulation of the antidepressant response operated by Negr-1, will be assessed by digital droplets PCR (ddPCR) and enzyme-linked immunosorbent assay (ELISA). The expression levels of the following genes involved in the NEGR-1 pathway will be tested in cerebrospinal fluid (CSF) cells. The genes include Abeta 1-42, tau, P-tau, MAPT, MAP2, GAP43, NCAM, SYP, VEGF, IGF-1, BDNF and FGF-2. Their expression levels will be tested in the CSF by Droplet Digital PCR (QX200 ddPCR BioRad), using Taqman Probes. Several housekeeping genes will be used for normalization. Biological samples will be processed by the laboratory of neurodegenerative and demyelinating diseases of the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico. Neuroimaging scans will be collected from MDD patients, BD patients and healthy controls at T0, and for MDD and BD patients at T1. The scans of neuroimaging will be performed using a 3-Tesla Philips Achieva MRI scanner and with an MRI-compatible EEG system). The investigators will collect data resting-state, at baseline and after 4 weeks of follow-up. The administration of drug therapy with venlafaxine (IMP of study) in MDD patients will be done according to normal clinical practice, following the indications in the CPR, the package insert and following medical prescription based on the clinical evaluation. The intervention study is related to the extra standard of care MRI that the MDD and BD patients will perform at baseline and after 4 weeks and to the cerebrospinal fluid collection (an invasive procedure not included in clinical practice for the management of these patients).

ELIGIBILITY:
Inclusion Criteria:

* GRUPPO 1: Recently diagnosed MDD, ongoing depressive episode, as determined by SCID-CV;
* Clinical indication to switch from current antidepressant therapy to venlafaxine due to lack of efficacy and/or tolerance and/or compliance.

GRUPPO 2: Recent diagnosis of BD with a current depressive episode, as determined by SCID-CV;

- absence of antidepressants in the patient's drug regimen.

GRUPPO 3: No diagnosis of psychiatric disorders made as a result of SCID-CV.

Exclusion Criteria:

* GRUPPO 1: - treatment with venlafaxine ongoing or within 6 months before the recruitment
* concomitant treatment with an irreversible MonoAmine Oxidase Inhibitor (I-MAO) or interruption of the IMAO treatment before 14 days from the recruitment;
* pregnant and breastfeeding woman;
* Lifetime comorbidity for psychotic disorders, as determined by the SCID-CV;
* Lifetime or recent history of suicide attempts or suicide-related behaviors and ideation (lifetime and/or recent C-SSRS Ideation or Behavior sub-score >0);
* Current, clinically meaningful, substance use disorders;
* Current comorbidity with neurological conditions or severe head trauma; -Neuropsychological diagnosis of intellectual disability;
* Presence of contraindications to lumbar puncture or MRI
* known hypersensitivity to the active substance venlafaxine or to any of the excipients
* Women of Childbearing Potential without a negative pregnancy test and not undertaking a high effective anticonception treatment at the recruitment

GRUPPO 2:

* Lifetime comorbidity for psychotic disorders, as determined by the SCID-CV;
* Current, clinically meaningful, substance use disorders;
* Current comorbidity with neurological conditions or severe head trauma;
* Neuropsychological diagnosis of intellectual disability;
* Presence of contraindications to lumbar puncture or MRI.

GRUPPO 3:

* Current or previous lifetime therapy with antidepressants
* Current, clinically meaningful, substance use disorders;
* Current comorbidity with neurological conditions or severe head trauma;
* Neuropsychological diagnosis of intellectual disability;
* Presence of contraindications to MRI scan

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
evaluate if venlafaxine induced a change in Negr1 gene expression in the whole blood of venlafaxine-treated MDD patients compared to antidepressant-free BD patients experiencing a depressive episode. | 4 weeks
  To observe a significant (p<0.05 at t test for continuous variable) differential concentration of Negr1 transcript (mRNA) and protein withing the T0 and T1 (4 weeks) in MDD patients treated with venlafaxine, respect to the antidepressant-free BD patient. The differential expression of Negr1 will be calculated for both patients' groups (MDD and BD) as the absolute variation between the blood Negr1 mRNA and plasmatic protein concentration measured at T0 and T1.

SECONDARY OUTCOMES:
To test the hypothesis that venlafaxine improves resting state brain connectivity in MDD patients through the modulation of Negr1 pathway, compared to venlafaxine-free BD patients | 4 weeks
  To observe a reorganization of beta-band functional connectivity in EEG-fMRI resting state recordings in MDD patients receiving venlafaxine for 4 weeks, compared to BD patients.
  - To establish a correlation between changes in EEG-FMRI connectivity metrics and Negr1 protein and/or transcript concentration.
To evaluate the variation of molecules able to modulate Negr1 gene expression or participating in Negr1 pathway between BD and MDD groups and within each single group over the follow-up period | 4 weeks
  Quantification of the blood differential concentrations of the ncRNAs BC048612 and miR-203 and of the Negr-1 related proteins Abeta 1-42, tau, P-tau, MAPT, MAP2, GAP43, NCAM, SYP, VEGF, IGF-1, BDNF, FGF-2 for each study group over the follow-up and To compare the differential concentration of the above markers between BD and MDD groups over the follow up period
To identify blood-based biomarkers of MDD | 4 weeks
  To compare peripheral (whole blood) expression levels of Negr1 and related proteins (Abeta 1-42, tau, P-tau, MAPT, MAP2, GAP43, NCAM, SYP, VEGF, IGF-1, BDNF, FGF-2) between HC, MDD, and BD patients.
To identify neuroimaging biomarkers of MDD | 4 weeks
  To compare beta-band functional connectivity from EEG-fMRI between HC, MDD, and BD patients.
To cross-sectionally assess the correspondence between central (CSF) and peripheral (whole blood) expression levels of Negr1 and related gene within MDD and BD groups at the baseline. | 4 weeks
  To quantify levels of Negr1 protein and transcript (mRNA) and of the Negr-1 related proteins Abeta 1-42, tau, P-tau, MAPT, MAP2, GAP43, NCAM, SYP, VEGF, IGF-1, BDNF, FGF-2 in the CSF of BD and MDD subjects at the baseline;
  - To correlate the CSF with the peripheral blood levels of these markers within BD and MDD group

CONTACTS AND LOCATIONS:
Overall Officials: Giandomenico Schiena, Doctor, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barreto RA, Walker FR, Dunkley PR, Day TA, Smith DW. Fluoxetine prevents development of an early stress-related molecular signature in the rat infralimbic medial prefrontal cortex. Implications for depression? BMC Neurosci. 2012 Oct 18;13:125. doi: 10.1186/1471-2202-13-125. PMID 23075086
- [Background] Brakowski J, Spinelli S, Dorig N, Bosch OG, Manoliu A, Holtforth MG, Seifritz E. Resting state brain network function in major depression - Depression symptomatology, antidepressant treatment effects, future research. J Psychiatr Res. 2017 Sep;92:147-159. doi: 10.1016/j.jpsychires.2017.04.007. Epub 2017 Apr 24. PMID 28458140
- [Background] Braun U, Schaefer A, Betzel RF, Tost H, Meyer-Lindenberg A, Bassett DS. From Maps to Multi-dimensional Network Mechanisms of Mental Disorders. Neuron. 2018 Jan 3;97(1):14-31. doi: 10.1016/j.neuron.2017.11.007. PMID 29301099
- [Background] Bromet EJ, Nock MK, Saha S, Lim CCW, Aguilar-Gaxiola S, Al-Hamzawi A, Alonso J, Borges G, Bruffaerts R, Degenhardt L, de Girolamo G, de Jonge P, Florescu S, Gureje O, Haro JM, He Y, Hu C, Karam EG, Kovess-Masfety V, Lee S, Lepine JP, Mneimneh Z, Navarro-Mateu F, Ojagbemi A, Posada-Villa J, Sampson NA, Scott KM, Stagnaro JC, Viana MC, Xavier M, Kessler RC, McGrath JJ; World Health Organization World Mental Health Survey Collaborators. Association Between Psychotic Experiences and Subsequent Suicidal Thoughts and Behaviors: A Cross-National Analysis From the World Health Organization World Mental Health Surveys. JAMA Psychiatry. 2017 Nov 1;74(11):1136-1144. doi: 10.1001/jamapsychiatry.2017.2647. PMID 28854302
- [Background] Brown EC, Clark DL, Hassel S, MacQueen G, Ramasubbu R. Thalamocortical connectivity in major depressive disorder. J Affect Disord. 2017 Aug 1;217:125-131. doi: 10.1016/j.jad.2017.04.004. Epub 2017 Apr 5. PMID 28407555
- [Background] Brunello N, Mendlewicz J, Kasper S, Leonard B, Montgomery S, Nelson J, Paykel E, Versiani M, Racagni G. The role of noradrenaline and selective noradrenaline reuptake inhibition in depression. Eur Neuropsychopharmacol. 2002 Oct;12(5):461-75. doi: 10.1016/s0924-977x(02)00057-3. PMID 12208564
- [Background] Burns DD, Spangler DL. Does psychotherapy homework lead to improvements in depression in cognitive-behavioral therapy or does improvement lead to increased homework compliance? J Consult Clin Psychol. 2000 Feb;68(1):46-56. doi: 10.1037//0022-006x.68.1.46. PMID 10710839
- [Background] Mayberg HS, Liotti M, Brannan SK, McGinnis S, Mahurin RK, Jerabek PA, Silva JA, Tekell JL, Martin CC, Lancaster JL, Fox PT. Reciprocal limbic-cortical function and negative mood: converging PET findings in depression and normal sadness. Am J Psychiatry. 1999 May;156(5):675-82. doi: 10.1176/ajp.156.5.675. PMID 10327898
- [Background] Cederquist GY, Asciolla JJ, Tchieu J, Walsh RM, Cornacchia D, Resh MD, Studer L. Specification of positional identity in forebrain organoids. Nat Biotechnol. 2019 Apr;37(4):436-444. doi: 10.1038/s41587-019-0085-3. Epub 2019 Apr 1. PMID 30936566
- [Background] Collins AL, Sullivan PF. Genome-wide association studies in psychiatry: what have we learned? Br J Psychiatry. 2013 Jan;202(1):1-4. doi: 10.1192/bjp.bp.112.117002. PMID 23284144
- [Background] Cross-Disorder Group of the Psychiatric Genomics Consortium; Lee SH, Ripke S, Neale BM, Faraone SV, Purcell SM, Perlis RH, Mowry BJ, Thapar A, Goddard ME, Witte JS, Absher D, Agartz I, Akil H, Amin F, Andreassen OA, Anjorin A, Anney R, Anttila V, Arking DE, Asherson P, Azevedo MH, Backlund L, Badner JA, Bailey AJ, Banaschewski T, Barchas JD, Barnes MR, Barrett TB, Bass N, Battaglia A, Bauer M, Bayes M, Bellivier F, Bergen SE, Berrettini W, Betancur C, Bettecken T, Biederman J, Binder EB, Black DW, Blackwood DH, Bloss CS, Boehnke M, Boomsma DI, Breen G, Breuer R, Bruggeman R, Cormican P, Buccola NG, Buitelaar JK, Bunney WE, Buxbaum JD, Byerley WF, Byrne EM, Caesar S, Cahn W, Cantor RM, Casas M, Chakravarti A, Chambert K, Choudhury K, Cichon S, Cloninger CR, Collier DA, Cook EH, Coon H, Cormand B, Corvin A, Coryell WH, Craig DW, Craig IW, Crosbie J, Cuccaro ML, Curtis D, Czamara D, Datta S, Dawson G, Day R, De Geus EJ, Degenhardt F, Djurovic S, Donohoe GJ, Doyle AE, Duan J, Dudbridge F, Duketis E, Ebstein RP, Edenberg HJ, Elia J, Ennis S, Etain B, Fanous A, Farmer AE, Ferrier IN, Flickinger M, Fombonne E, Foroud T, Frank J, Franke B, Fraser C, Freedman R, Freimer NB, Freitag CM, Friedl M, Frisen L, Gallagher L, Gejman PV, Georgieva L, Gershon ES, Geschwind DH, Giegling I, Gill M, Gordon SD, Gordon-Smith K, Green EK, Greenwood TA, Grice DE, Gross M, Grozeva D, Guan W, Gurling H, De Haan L, Haines JL, Hakonarson H, Hallmayer J, Hamilton SP, Hamshere ML, Hansen TF, Hartmann AM, Hautzinger M, Heath AC, Henders AK, Herms S, Hickie IB, Hipolito M, Hoefels S, Holmans PA, Holsboer F, Hoogendijk WJ, Hottenga JJ, Hultman CM, Hus V, Ingason A, Ising M, Jamain S, Jones EG, Jones I, Jones L, Tzeng JY, Kahler AK, Kahn RS, Kandaswamy R, Keller MC, Kennedy JL, Kenny E, Kent L, Kim Y, Kirov GK, Klauck SM, Klei L, Knowles JA, Kohli MA, Koller DL, Konte B, Korszun A, Krabbendam L, Krasucki R, Kuntsi J, Kwan P, Landen M, Langstrom N, Lathrop M, Lawrence J, Lawson WB, Leboyer M, Ledbetter DH, Lee PH, Lencz T, Lesch KP, Levinson DF, Lewis CM, Li J, Lichtenstein P, Lieberman JA, Lin DY, Linszen DH, Liu C, Lohoff FW, Loo SK, Lord C, Lowe JK, Lucae S, MacIntyre DJ, Madden PA, Maestrini E, Magnusson PK, Mahon PB, Maier W, Malhotra AK, Mane SM, Martin CL, Martin NG, Mattheisen M, Matthews K, Mattingsdal M, McCarroll SA, McGhee KA, McGough JJ, McGrath PJ, McGuffin P, McInnis MG, McIntosh A, McKinney R, McLean AW, McMahon FJ, McMahon WM, McQuillin A, Medeiros H, Medland SE, Meier S, Melle I, Meng F, Meyer J, Middeldorp CM, Middleton L, Milanova V, Miranda A, Monaco AP, Montgomery GW, Moran JL, Moreno-De-Luca D, Morken G, Morris DW, Morrow EM, Moskvina V, Muglia P, Muhleisen TW, Muir WJ, Muller-Myhsok B, Murtha M, Myers RM, Myin-Germeys I, Neale MC, Nelson SF, Nievergelt CM, Nikolov I, Nimgaonkar V, Nolen WA, Nothen MM, Nurnberger JI, Nwulia EA, Nyholt DR, O'Dushlaine C, Oades RD, Olincy A, Oliveira G, Olsen L, Ophoff RA, Osby U, Owen MJ, Palotie A, Parr JR, Paterson AD, Pato CN, Pato MT, Penninx BW, Pergadia ML, Pericak-Vance MA, Pickard BS, Pimm J, Piven J, Posthuma D, Potash JB, Poustka F, Propping P, Puri V, Quested DJ, Quinn EM, Ramos-Quiroga JA, Rasmussen HB, Raychaudhuri S, Rehnstrom K, Reif A, Ribases M, Rice JP, Rietschel M, Roeder K, Roeyers H, Rossin L, Rothenberger A, Rouleau G, Ruderfer D, Rujescu D, Sanders AR, Sanders SJ, Santangelo SL, Sergeant JA, Schachar R, Schalling M, Schatzberg AF, Scheftner WA, Schellenberg GD, Scherer SW, Schork NJ, Schulze TG, Schumacher J, Schwarz M, Scolnick E, Scott LJ, Shi J, Shilling PD, Shyn SI, Silverman JM, Slager SL, Smalley SL, Smit JH, Smith EN, Sonuga-Barke EJ, St Clair D, State M, Steffens M, Steinhausen HC, Strauss JS, Strohmaier J, Stroup TS, Sutcliffe JS, Szatmari P, Szelinger S, Thirumalai S, Thompson RC, Todorov AA, Tozzi F, Treutlein J, Uhr M, van den Oord EJ, Van Grootheest G, Van Os J, Vicente AM, Vieland VJ, Vincent JB, Visscher PM, Walsh CA, Wassink TH, Watson SJ, Weissman MM, Werge T, Wienker TF, Wijsman EM, Willemsen G, Williams N, Willsey AJ, Witt SH, Xu W, Young AH, Yu TW, Zammit S, Zandi PP, Zhang P, Zitman FG, Zollner S, Devlin B, Kelsoe JR, Sklar P, Daly MJ, O'Donovan MC, Craddock N, Sullivan PF, Smoller JW, Kendler KS, Wray NR; International Inflammatory Bowel Disease Genetics Consortium (IIBDGC). Genetic relationship between five psychiatric disorders estimated from genome-wide SNPs. Nat Genet. 2013 Sep;45(9):984-94. doi: 10.1038/ng.2711. Epub 2013 Aug 11. PMID 23933821
- [Background] DeRubeis RJ, Hollon SD, Amsterdam JD, Shelton RC, Young PR, Salomon RM, O'Reardon JP, Lovett ML, Gladis MM, Brown LL, Gallop R. Cognitive therapy vs medications in the treatment of moderate to severe depression. Arch Gen Psychiatry. 2005 Apr;62(4):409-16. doi: 10.1001/archpsyc.62.4.409. PMID 15809408
- [Background] Dichter GS, Gibbs D, Smoski MJ. A systematic review of relations between resting-state functional-MRI and treatment response in major depressive disorder. J Affect Disord. 2015 Feb 1;172:8-17. doi: 10.1016/j.jad.2014.09.028. Epub 2014 Sep 26. PMID 25451389
- [Background] Disner SG, Beevers CG, Haigh EA, Beck AT. Neural mechanisms of the cognitive model of depression. Nat Rev Neurosci. 2011 Jul 6;12(8):467-77. doi: 10.1038/nrn3027. PMID 21731066
- [Background] Drevets WC, Price JL, Simpson JR Jr, Todd RD, Reich T, Vannier M, Raichle ME. Subgenual prefrontal cortex abnormalities in mood disorders. Nature. 1997 Apr 24;386(6627):824-7. doi: 10.1038/386824a0. PMID 9126739